CLINICAL TRIAL: NCT02307812
Title: Ramucirumab Use in Combination With Paclitaxel in Gastric or Gastroesophageal Junction Adenocarcinoma; Temporary Authorization for Use (ATU) in France
Status: Approved for marketing | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 15263; I4T-FR-JVCS (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-11-25; First posted 2014-12-04 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ramucirumab; Paclitaxel

INTERVENTIONS:
Drug: Ramucirumab — Administered intravenously (IV)
  Other Names: IMC-1121B; LY3009806
Drug: Paclitaxel — Administered IV

SUMMARY:
The treating physician/investigator contacts Lilly when, based on their medical opinion, a patient meets the criteria for inclusion in the ATU.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically or cytologically confirmed gastric adenocarcinoma, including gastroesophageal junction (GEJ) adenocarcinoma (Participants with adenocarcinoma of the distal esophagus are eligible if the primary tumor involves the GEJ.) after prior chemotherapy.
* Acceptable prior chemotherapy regimens for this protocol are combination chemotherapy regimens that include platinum or fluoropyrimidine components (acceptable prior platinum agents are cisplatin, carboplatin, or oxaliplatin; acceptable prior fluoropyrimidine agents are 5-fluorouracil (5-FU) and capecitabine). Prior trastuzumab use in human epidermal growth factor receptor 2 positive (HER2+) participants is accepted too.
* The participant is eligible for treatment by chemotherapy and has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.

Exclusion Criteria:

* Participant has a known allergy to any of the treatment components.

Sex: All
Age Groups: Child, Adult, Older Adult